CLINICAL TRIAL: NCT06911047
Title: Dementia Prevention Internet-Based Intervention: Randomized Controlled Trial and Knowledge Translation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study did not receive funding.
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Levinson_DCI
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Dementia Prevention
Keywords: web-based intervention; knowledge translation; clinical trial; education and training; alzheimer disease; caregiver; dementia; internet
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Participant
Masking Description: Efforts will be made to blind participants to their allocation group (intervention or control). To do this, we will ensure that promotional advertisements do not contain logos or direct website links. The informed consent form will not contain the exact outcome measures or the title of the intervention. To the best of our abilities, allocation concealment will be aided by referring to the intervention as 'e-learning about cognitive impairment and dementia prevention', without biasing participants to study hypotheses or study design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education Intervention (Experimental): Participants in the intervention group will be provided e-learning about dementia prevention and promoting brain health, consisting of following components:
  1. One multimedia e-learning lesson on promoting brain health and preventing dementia;
  2. A series of 12 'micro-learning' emails (3 emails/week) with small segments of content to reinforce the material from the lesson.
  3. Curated resources related to dementia risk factors
  Interventions: Behavioral: Education Intervention
- Education Control (Active Comparator): Participants in the control group will be provided e-learning about mild cognitive impairment, consisting of following components:
  1. One multimedia e-learning lesson on mild cognitive impairment;
  2. A series of 12 'micro-learning' emails (3 emails/week) with small segments of content to reinforce the material from the lesson.
  3. Curated resources related to mild cognitive impairment
  Interventions: Behavioral: Education Control

INTERVENTIONS:
Behavioral: Education Intervention — Participants in the intervention group will be provided e-learning about dementia prevention and promoting brain health, consisting of following components: 1. One multimedia e-learning lesson on promoting brain health and preventing dementia; 2. A series of 12 'micro-learning' emails (3 emails/week) with small segments of content to reinforce the material from the lesson. 3. Curated resources related to dementia risk factors
  Arms: Education Intervention
Behavioral: Education Control — Participants in the control group will be provided e-learning about mild cognitive impairment, consisting of following components: 1. One multimedia e-learning lesson on mild cognitive impairment; 2. A series of 12 'micro-learning' emails (3 emails/week) with small segments of content to reinforce the material from the lesson. 3. Curated resources related to mild cognitive impairment
  Arms: Education Control

SUMMARY:
In this proposal, the investigators plan to study the effectiveness of a web-based intervention on dementia prevention knowledge, intentions, and behaviour change related to dementia risk. Participants will be randomized to one of two groups - intervention and control. Participants randomized to the intervention group will receive the dementia prevention e-learning. Participants in the control group will be assigned an alternate-topic e-learning lesson. All participants will be given access to all e-learning at the conclusion of the study.

The purpose of this phase is to explore if and how our dementia prevention e-learning influences participants' knowledge, intentions and health behaviours related to dementia risk.

The investigators will also engage in participatory co-design with community partners using focus groups to determine pragmatic ways to effectively disseminate e-learning programs to support knowledge about dementia and preventative measures within equity-deserving groups.

DETAILED DESCRIPTION:
Background:

With our aging population, the prevalence of dementia is increasing dramatically. Developing a better understanding of how dementia can be prevented and sharing information about how Canadians can reduce their risk of developing dementia or delay its onset is critical to keeping Canadians healthy and improving quality of life. Web-based interventions in dementia have been shown to be effective for a range of outcomes, but very few have been widely implemented or rigorously studied; additionally, national, and provincial guidelines have all highlighted the importance of online resources to improve dementia prevention education. This has been further brought into focus by the coronavirus pandemic. While there have been studies of web-based health information on intentions and behaviour change, the vast majority of those studies have looked at text-based health information, rather than internet-based interventions that have incorporated best practices in instructional design for e-learning. The investigators developed a high-quality, award-winning web- and email-based dementia prevention education platform for care partners, which includes asynchronous, multimedia e-learning lessons and email-based 'micro-learning' content to reinforce the learning. The investigators recently conducted a Randomized Controlled Trial (RCT) of an internet-based, multi-media, instructionally designed dementia prevention intervention (DementiaRisk) in Canadian adults without a diagnosis of dementia. Results, which are currently being prepared for publication, showed that the DementiaRisk resource improved knowledge, intentions to engage in healthy behaviours, and health behaviours related to dementia risk reduction, and was positively rated and well accepted by participants. This resource is now publicly accessible at DementiaRisk.ca.

However, we know that people who live in poverty are more likely to develop dementia compared to people of higher socioeconomic status. Lower level of education in childhood is a known risk factor for dementia, but there are many other social determinants of health (e.g., income, employment, housing, and others) that may impact knowledge and behaviours related to dementia risk or protective factors. A range of positive effects have been shown for web-based interventions for various target audiences (e.g., health care providers and family/friend care partners), on a wide range of outcomes (e.g., knowledge, attitudes, burden, stress, and others). Interventions delivered through the web also allow for greater accessibility to a multitude of users, facilitating scale and spread. We therefore wish to study the impact of the DementiaRisk resource in a new equity-deserving population.

Objective:

In this proposal, the investigators plan to study the effectiveness of our web-based intervention on dementia prevention knowledge, intentions, and behaviour change.

Methods:

Design, Setting, and Participants:

This study is a sequential explanatory mixed methods design randomized controlled trial. Following eligibility screening, informed consent, and baseline socio-demographic measures, participants will be randomized either to the intervention group or the control group. Those adults (age ≥ 16) who have no prior diagnosis of dementia, have internet and email access, and are fluent in English will be eligible to participate in the RCT. Participants will be randomized and directed to their assigned learning path after submitting online informed consent and baseline measures using the Division of e-Learning Innovation's research platform. Participants will be randomized using a block randomization. To the best of our ability, efforts will be made to blind participants to their allocation group and study hypotheses.

Focus groups will be conducted with 6-10 representative participants (not involved in the RCT) including: intervention agents/organization staff and leaders, people who identify as low income, people who identify as family/friend care partners of people living with dementia, and/or people living with dementia.

Intervention:

Participants randomized to the intervention group will receive the dementia prevention e-learning. Participants in the control group will be assigned an alternate-topic e-learning lesson. All participants will be given access to all e-learning at the conclusion of the study.

Focus groups will use an interview guide informed by the CFIR Framework.

Outcomes:

The purpose of this phase is to explore if and how our dementia prevention e-learning influences participants' knowledge, intentions and health behaviours related to dementia risk.

The specific aims are:

1. To evaluate whether exposure to the e-learning intervention changes knowledge of dementia risk factors, intention to engage in risk reduction activities, and health behaviours related to dementia prevention.
2. To explore qualitative aspects such as participants' engagement and satisfaction with the intervention, as well as barriers and facilitators to use, through surveys and synchronous online focus groups.

Focus groups will focus on better understanding barriers and facilitators for uptake, use, and dissemination of e-learning within a lower-income setting.

Implications and Relevance:

The results of this study will contribute to the planning of a larger randomized controlled trial (RCT) in the future; as well as the evaluation of innovative, cost-effective, and efficient dementia prevention resources that can complement traditional approaches. The intervention could be easily scaled and spread to complement other dementia education methods. Focus groups will help to inform further implementation and scale and spread to disadvantaged populations.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:
* No prior diagnosis of dementia
* Live in Canada
* 16 years of age and over
* Good command of the English language
* Access to email and internet
* Comfortable using email and internet, and
* Ability to grant online informed consent

Exclusion Criteria:

* Prior diagnosis of dementia
* Lives outside of Canada
* Not 16 years of age or over
* Does not speak English,
* Does not have access to email or internet
* Is not comfortable using email of internet
* Does not grant informed consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-01-29 (Actual); Study Completion 2026-01-29 (Actual)

PRIMARY OUTCOMES:
1. Knowledge change (custom 15-item knowledge questionnaire related to key dementia prevention modifiable risk factors | 0 weeks, 4 weeks, 12 weeks
  A custom 15-item knowledge questionnaire (multiple true-false response) to measure change related to key dementia prevention modifiable risk factors. Items are pulled from other validated surveys (i.e., Dementia Knowledge Assessment Scale) and key dementia prevention modifiable risk factors.

SECONDARY OUTCOMES:
Intentions change (custom 10-item intentions questionnaire related to key dementia prevention modifiable risk factors) | 0 weeks, 4 weeks, 12 weeks
  Intentions related to dementia prevention. A custom 10-item intentions questionnaire (7 point Likert scale) to measure intentions to change related to key dementia prevention modifiable risk factors. Items were created based on key modifiable risk factors related to dementia as identified by the 2020 Lancet Commission Report.
Behaviour change related to dementia prevention (custom 42-item health behaviours questionnaire) | 0 weeks, 4 weeks, 12 weeks
  Behaviour change related to dementia prevention. A custom 42-item health behaviours questionnaire (Likert response options) to measure health behaviours related to key dementia prevention modifiable risk factors. Items are pulled from other validated surveys (Health and Behaviour Survey, Godin Leisure Time Exercise Questionnaire, World Health Organization for smoking status, etc.) and key dementia prevention modifiable risk factors.

OTHER OUTCOMES:
Intervention adherence (time spent) | 4 weeks
  Lesson completion data, email open rates, and resource downloads will be collected and saved to quantify the time(s) spent on intervention activities.
Participant satisfaction | 4 weeks
  A custom satisfaction questionnaire data adapted from the Information Assessment Method For All (IAM4all) will be collected and saved to assess satisfaction with the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No